CLINICAL TRIAL: NCT07373210
Title: Conditioning, Open-label Placebo for Pain Management in Adolescents and Young Adults Undergoing Bernese Periacetabular Osteotomy (PAO)
Brief Title: Open-label Placebo for Pain Management in Adolescents and Young Adults Undergoing Bernese Periacetabular Osteotomy
Acronym: COLP PAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-44743
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Periacetabular Osteotomy; Opiates
Keywords: periacetabular osteotomy; opiates
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-label Placebo (COLP) (Experimental): One placebo tablet will be taken with each oral opioid dose, 5mg Oxycodone, 3 times per day, beginning on post-operative day 1.
  Interventions: Other: Open-Label Placebo; Other: Treatment as usual
- Treatment As Usual (TAU) (Experimental): Treatment As Usual (TAU) participants will receive their standard opioid dose, 5mg Oxycodone pill, three times a day beginning on post-operative day 1.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Open-Label Placebo — One placebo tablet will be taken with each oral opioid dose, 5mg Oxycodone, 3 times per day, beginning on post-operative day 1.
  Arms: Open-label Placebo (COLP)
Other: Treatment as usual — Treatment As Usual (TAU) participants will receive their standard opioid dose, 5mg Oxycodone pill, three times a day beginning on post-operative day 1.

SUMMARY:
In this randomized controlled trial, 64 participants undergoing PAO at UCSF will be enrolled and randomized to receive either COLP plus treatment as usual (TAU) or TAU alone. Patients in the COLP arm will receive placebo pills alongside prescribed opioids and at scheduled intervals, beginning on postoperative day one. Weekly follow-up will be conducted for six weeks postoperatively via remote surveys and video visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 to 40 years old, and
* Undergo primary Bernese Periacetabular osteotomy (PAO) for symptomatic developmental dysplasia of the hip (DDH), and
* Opioid-naïve prior to operation, and
* Capable of completing study procedures, including daily pain and medication diaries as well as weekly questionnaires.

Exclusion Criteria:

* Undergoing PAO revision or any concurrent major surgical procedure
* History of opioid use, substance use disorders, or alcohol abuse
* Those with cognitive or physical impairments that would interfere with providing their own consent and the completion of study-related tasks
* Pregnant individuals or those planning to become pregnant during the study period

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Conditioning + Open-Label Placebo (COLP) results in significantly reduced opioid consumption compared with Treatment as Usual (TAU) | Admission to 6 weeks post-operatively
  COLP participants will take one placebo pill with their standard post-operative medications. TAU participants will take standard post-operative medications. Opioid Daily Diary and surveys will compare the opioid amount.
To determine if 6 weeks of COLP results in reduced pain perception compared with TAU. | Admission to 6 weeks post-operatively.
  Pain perception will be measured by surveys.

SECONDARY OUTCOMES:
Duration of time in days following surgery until patients establish independence with physical therapy | Post-operative Day 1 to 6 weeks.
  Participants will be treated by physical therapy services after surgery until their physical therapist determines that services are no longer needed.
Length of hospital stay | Admission to discharge, up to 6 weeks
  Participants will be admitted to the hospital following surgery until cleared for discharge.
Time to return to school or work | Discharge to first day of school or work, up to 6 weeks post-operatively
  Participants will be asked to record date they have returned to school or work after surgery. The amount of time it takes to return, may determine if they are struggling with pain.
Urinary retention | During hospitalization, until discharge, up to 6 weeks
  Participants will be assessed in hospital to determine whether or not they experience urinary retention post surgery, a potential side effect of opioid consumption.
Constipation & First Bowel Movement | Post-operatively to first flatus and bowel movement, up to 6 weeks
  Participants will record the first time they flatulate, the number of days until their first bowel movement after surgery to assess constipation, a potential side effect of opioid consumption.
Number of postoperative clinical contacts in COLP compared to TAU | Post-operatively to 6 weeks
  The number of interactions or communication between the participant and medical providers. This includes follow-up visits, phone calls, or messages.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Diab, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furie KS, James K, Kaptchuk TJ, Diab M. Effectiveness of conditioning + open-label placebo for post-operative pain management in adolescent idiopathic scoliosis. Pain Manag. 2025 Jul;15(7):363-371. doi: 10.1080/17581869.2025.2520148. Epub 2025 Jun 19. PMID 40536435
- [Background] Carvalho C, Caetano JM, Cunha L, Rebouta P, Kaptchuk TJ, Kirsch I. Open-label placebo treatment in chronic low back pain: a randomized controlled trial. Pain. 2016 Dec;157(12):2766-2772. doi: 10.1097/j.pain.0000000000000700. PMID 27755279
- [Background] Blease C, Colloca L, Kaptchuk TJ. Are open-Label Placebos Ethical? Informed Consent and Ethical Equivocations. Bioethics. 2016 Jul;30(6):407-14. doi: 10.1111/bioe.12245. Epub 2016 Feb 3. PMID 26840547
- [Background] von Wernsdorff M, Loef M, Tuschen-Caffier B, Schmidt S. Effects of open-label placebos in clinical trials: a systematic review and meta-analysis. Sci Rep. 2021 Feb 16;11(1):3855. doi: 10.1038/s41598-021-83148-6. PMID 33594150
- [Background] Kirchhof J, Petrakova L, Brinkhoff A, Benson S, Schmidt J, Unteroberdorster M, Wilde B, Kaptchuk TJ, Witzke O, Schedlowski M. Learned immunosuppressive placebo responses in renal transplant patients. Proc Natl Acad Sci U S A. 2018 Apr 17;115(16):4223-4227. doi: 10.1073/pnas.1720548115. Epub 2018 Apr 2. PMID 29610294
- [Background] Ader R, Mercurio MG, Walton J, James D, Davis M, Ojha V, Kimball AB, Fiorentino D. Conditioned pharmacotherapeutic effects: a preliminary study. Psychosom Med. 2010 Feb;72(2):192-7. doi: 10.1097/PSY.0b013e3181cbd38b. Epub 2009 Dec 22. PMID 20028830
- [Background] Doering BK, Rief W. Utilizing placebo mechanisms for dose reduction in pharmacotherapy. Trends Pharmacol Sci. 2012 Mar;33(3):165-72. doi: 10.1016/j.tips.2011.12.001. Epub 2012 Jan 25. PMID 22284159
- [Background] Sandler AD, Glesne CE, Bodfish JW. Conditioned placebo dose reduction: a new treatment in attention-deficit hyperactivity disorder? J Dev Behav Pediatr. 2010 Jun;31(5):369-75. doi: 10.1097/DBP.0b013e3181e121ed. PMID 20495473
- [Background] Nurko S, Saps M, Kossowsky J, Zion SR, Di Lorenzo C, Vaz K, Hawthorne K, Wu R, Ciciora S, Rosen JM, Kaptchuk TJ, Kelley JM. Effect of Open-label Placebo on Children and Adolescents With Functional Abdominal Pain or Irritable Bowel Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):349-356. doi: 10.1001/jamapediatrics.2021.5750. PMID 35099543
- [Background] Flowers KM, Patton ME, Hruschak VJ, Fields KG, Schwartz E, Zeballos J, Kang JD, Edwards RR, Kaptchuk TJ, Schreiber KL. Conditioned open-label placebo for opioid reduction after spine surgery: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1828-1839. doi: 10.1097/j.pain.0000000000002185. PMID 33449503